CLINICAL TRIAL: NCT05876858
Title: EXPLORER Total Body PET/CT Imaging for Myofascial Pain
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1834390; 1R61AT012187-01 (NIH)
Record Dates: First submitted 2023-04-27; First posted 2023-05-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Pain
Keywords: total body positron emission tomography
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Participants will undergo two PET/CT scans with two different radiotracers. In addition, participants will complete questionnaires to establish the association of quantitative TB-PET/CT measures with the NIH Helping to End Addiction Long-term (HEAL) outcome measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET/CT scans (Experimental): Each subject will undergo a dynamic 18F-FDG PET/CT scan and a dynamic 11C-butanol PET/CT scan on the EXPLORER total-body PET/CT system
  Interventions: Drug: 18F-FDG; Drug: 11C-butanol

INTERVENTIONS:
Drug: 18F-FDG — Each subject will undergo a dynamic 18F-FDG PET/CT scan (this drug is FDA approved) and a dynamic 11C-butanol PET/CT scan (this drug is under an IND) on the EXPLORER total-body PET/CT system. The two scans will be performed on the same day or within a period of up to four weeks depending on subject, imaging agent and scanner availability. Subjects will be asked to complete the HEAL questionnaires before or after their PET/CT scan on each day.
Drug: 11C-butanol — Each subject will undergo a dynamic 18F-FDG PET/CT scan (this drug is FDA approved) and a dynamic 11C-butanol PET/CT scan (this drug is under an IND) on the EXPLORER total-body PET/CT system. The two scans will be performed on the same day or within a period of up to four weeks depending on subject, imaging agent and scanner availability. Subjects will be asked to complete the HEAL questionnaires before or after their PET/CT scan on each day.

SUMMARY:
The main objective of this study is to establish novel measures derived from Total-body-Positron Emission Tomography/Computed Tomography (TB-PET/CT) as quantitative biomarkers for the investigation of myofascial pain. The TB-PET/CT assessed measures are those reflective of myofascial tissue metabolism, perfusion, and fatty infiltration.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a prevalent and debilitating condition representing a significant societal burden. It is a chronic muscular pain disorder involving one muscle or groups of muscles, which is frequently accompanied by decreased range of motion, weakness, autonomic phenomena, depression, anxiety, sleep disturbance, and altered mental function. MPS affects up to 85% of patients with chronic pain and it is one of the most frequent reasons for referral to large pain clinics. The highest age-specific incidence rate is in the early 20's while prevalence increases with age until the sixth decade of life. This specific epidemiology of the disease creates a large economic burden on society due to not only health-care related expense but, especially, due to disabilities and work absenteeism.

Patients often receive treatment for myofascial pain, which are often neither standardized nor evidence-based. Treatment for myofascial pain consists of pharmacologic and nonpharmacologic interventions. Pharmacologic therapies include nonsteroidal anti-inflammatory drugs, muscle relaxants, benzodiazepines, and opioids. All these therapies have systemic physical side effects which can lead to severe chronic complications, especially when chronically prescribed. All of these are also known as being addictive or misused/overused. Non-pharmaceutical approaches ranging from non-invasive physical force-based manipulations to mini-invasive interventions such as acupuncture. These non-pharmacologic approaches are associated with minimal or negligible side effects and have been recently introduced into a conceptual model of integrative medicine.

There are no validated biomarkers for qualitative or quantitative assessment of MPS, which can be used to guide clinical management. It is crucial to have a reliable biomarker to assess therapy or intervention response. While many approaches have been attempted with several different techniques including MRI and US, there has not been a solid effort to assess a functional/molecular biomarker with PET/CT. Conventional PET/CT scanners are affected by low signal efficiency collection and low spatial resolution, which have made them unpractical to develop MPS biomarkers. However, the first Total Body PET/CT (TB-PET/CT) was successful in imaging the whole body simultaneously (field of view of 194 cm), with low injected activity doses (1/20 of the regular dose) and reduced acquisition times (less than 1 minute). The Investigators conducted several first-in-human studies using the TB-PET/CT system in participants with cancer, autoimmune arthritis, Covid-19, neurodegeneration and HIV. This included imaging the entire body down to a single nail of the finger. These strong data clearly address challenges of current PET/CT systems, such as their inability to assess the entire body in the same phase of radiotracer uptake, long scan times resulting from sequential acquisitions of the entire body that may not be well-tolerated by patients, significant ionizing radiation exposure in the context of monitoring chronic disease activity in a longitudinal setting, and limited PET spatial resolution for measuring radiotracer uptake in small lesions. Therefore, TB-PET/CT is poised to shift the paradigm in a range of research areas towards utilizing of advanced imaging technology. The PET radiotracer Fluorodeoxyglucose (18F-FDG) is a marker of glucose metabolism and is the mostly common radiotracer used in the PET imaging field. This radiotracer is FDA approved. 11C-Butanol is a marker for blood perfusion. This radiotracer is not FDA approved, and it will be used under an IND for this study. In summary, these observations support our overall scientific premise that total body PET/CT can be used in the assessment of myofascial tissue dysfunction using both FDG and 11C-Butanol.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign an informed consent form
* Ability to adhere to the study visit schedule and all protocol requirements.
* Men and women ≥18 years of age
* Current self-report of chronic low back pain (cLBP) which has persisted for the past 3 months AND has resulted in pain on > 50% of days in the past 6 months
* At least one palpable nodule or taut band in paraspinal, quadratus lumborum, or gluteal muscles
* Reproduction of the patient's dominant pain with palpation of a muscle nodule or taut band
* Predominantly paramedian pain (may be uni-lateral or bi-lateral)
* Willing and able to lay motionless in a supine position on 2 different occasions:

  * 60-70 minutes 18F-FDG scan
  * 10-20 minutes 11C-Butanol Scan
* Willing and able to fast for at least 6 hours before and for the duration of the scan
* Willing to avoid strenuous exercise for 24 hours before the scan visit

Exclusion Criteria:

* No Primary Care Physician
* History of any cancer (except non-melanoma skin cancer)
* History of spine infection (discitis or osteomyelitis) or spine tumor
* History of ankylosing spondylitis, rheumatoid arthritis, polymyalgia rheumatica, psoriatic arthritis, or lupus or other connective tissue diseases.
* Confounding conditions that are known to be responsible for inducing pain
* Implants at or in the region of the sites of interest
* Diagnosis of any vertebral fracture in the last 6 months
* Cauda equina syndrome or lumbar radiculopathy with functional motor deficit (strength<4/5 on manual motor testing)
* Spinal implants (including fixation hardware, spinal cord stimulator, intra-thecal pumps)
* Predominantly central pain
* Pain below the knee
* Positive straight leg raise test
* Symptomatic hip arthritis
* Fasting blood glucose level greater than 200 mg/dl before administration of 18F-FDG
* Self-reported history of dysphoria or anxiety in closed spaces
* Pregnant or lactating subjects
* Body weight more than 240 kg (529 pounds) due to the weight limitation of the scanner bed
* Prisoners
* Inability to speak, read, and write in the English language
* Concurrent or prior enrollment in a separate research study involving a PET scan performed within the last 12 months for research purposes only
* Any other criteria, which would make the subject unsuitable to participate in this study as determined by the Principal Investigator (e.g., subject has a Legally Authorized Representative and cannot consent for him/herself)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
HEAL outcome measure | This is a cross-sectional study and the PEG score will be evaluated at baseline on the day of the scans.
  Our primary outcome measure is the NIH Helping to End Addiction Long-term (HEAL) measure: PEG (Pain, Enjoyment, General Activity) score, which quantitatively evaluates pain intensity and interference. This is a score from 0 to 10.
Differentiate Myofascial tissues | Baseline; Up to 30 minutes (30 min being the time to fil out questionnaires)
  The primary outcome measure is the Standardized Uptake Value (SUV) derived from the Positron Emission Tomography scans. This is a unitless quantity.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Nardo, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No